CLINICAL TRIAL: NCT05083676
Title: A Study Protocol on Peer Digital Acceset (PDA): A Randomized Controlled Trial to Translate Online Peer Support for Youth Mental Well-being
Brief Title: A Study Protocol on Peer Digital Acceset (PDA)
Acronym: PDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The N.1 Institute for Health (N.1) (Other)
Collaborators: Acceset (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Acceset Prospective Study
Record Dates: First submitted 2021-09-15; First posted 2021-10-19 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Issue
Keywords: Mattering; Self-hood; Compassion; Mindfulness; Digital Peer Support Intervention; peer emotional disclosure; community; Mental Well-being; Digital biomarkers
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We propose an interventional prospective study with hybrid design that evaluates both implementation of Acceset platform (e.g., fidelity, adoption, and utility), as well as clinical outcomes (e.g., anxiety and depressive symptoms) using randomized controlled trials. The intervention comprises of two components: (1) digital peer support training and (2) digital intervention involving three features, specifically emotionality, motivations and functional improvement serving as digital markers of psychological well-being, the peer emotional disclosure process, as well as community engagement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceset Intervention (Experimental): The qualified participants (seekers) will be randomly allocated into two arms. Arm 1 (n = 50) seekers will engage with the Acceset platform for a period of 3 weeks, together with befrienders (n = 30) and moderators (n = 30). Both seekers and befrienders will be monitored using a questionnaire battery listed (including help seeking behaviors beyond the Acceset platform) at 4 time points: baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects).
  Interventions: Behavioral: Acceset Intervention
- waitlist for Acceset intervention (Active Comparator): Arm 2 (n = 50) a control group will be placed on a waitlist for Acceset intervention. These individuals will be age and gender matched with the intervention group (i.e., arm 1). Their mental well-being, as well as their help seeking behavior, at the same time points and via the same questionnaire battery will be compared with those in arm 1.
  Interventions: Behavioral: Acceset Intervention

INTERVENTIONS:
Behavioral: Acceset Intervention — . The intervention comprises of: i) Digital peer support training for youth befrienders to equip them with the knowledge and application of the four active ingredients-Mattering, selfhood, compassion, and mindfulness-to provide effective peer support as they respond to youth seekers' emotional experiences.
  ii) Acceset Intervention with features or digital markers of psychological well-being, peer emotional disclosure process and community engagement.
  Other Names: Digital Peer Support Intervention

SUMMARY:
This protocol delineates a randomized controlled trial for evaluating the implementation and clinical effectiveness of Assecet, a digital peer support intervention for youth mental well-being, which comprises two components. The digital peer support training curriculum aims to equip youth befrienders (i.e., peers who provide support) with knowledge and skills in harnessing four active ingredients of youth mental well-being-specifically, Mattering, selfhood, compassion, and mindfulness, in providing effective peer support for seekers (peers who seek support). The Acceset intervention that involves three components-digital biomarkers of psychological well-being, peer emotional disclosure process and community engagement.

DETAILED DESCRIPTION:
Background: The burgeoning mental health issues among emerging adults (ages 19 to 25) worldwide has fuelled concerns about youths' widespread experiences of emotional distress, specifically concerning anxiety and depression, and coping mechanisms. Digital peer support intervention has demonstrated varying degrees of clinical effectiveness for positive health and psychological outcomes across different developmental stages. The onset of the COVID-19 pandemic has resulted in prolonged isolation and reduced social connections, and emerging literature is amounting to the import of digital peer emotional disclosure and support for young people psychological well-being. However, much remains to be explored regarding implementation and clinical effectiveness-how best to conduct digital peer intervention in support of youths' psychological well-being, and the associated mechanism of change.

Objective: This protocol delineates a randomized controlled trial for evaluating the implementation and clinical effectiveness of Assecet, a digital peer support intervention for youth mental well-being, which comprises two components. The digital peer support training curriculum aims to equip youth befrienders (i.e., peers who provide support) with knowledge and skills in harnessing four active ingredients of youth mental well-being-specifically, Mattering, selfhood, compassion, and mindfulness, in providing effective peer support for seekers (peers who seek support). The Acceset intervention that involves three components-digital biomarkers of psychological well-being, peer emotional disclosure process and community engagement.

Methods: Participants will consist of 100 students ages 19 to 25 from the National University of Singapore to engage with the Acceset platform. At the time of recruitment, individuals will be screened for inclusion and exclusion criteria based on self-reporting. The qualified participants (seekers) will be randomly allocated into two arms. Arm 1 (n = 50) seekers will engage with the Acceset platform for a period of 3 weeks, together with befrienders (n = 30) and moderators (n = 30). Arm 2 (n = 50) a control group will be placed on a waitlist for Acceset intervention. These individuals will be age and gender matched with the intervention group (i.e., arm 1). Their mental well-being, as well as their help seeking behavior, at the same time points and via the same questionnaire battery will be compared with those in arm 1. Both seekers and befrienders will be monitored using a questionnaire battery listed (including help seeking behaviors beyond the Acceset platform) at 4 time points: baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects). The implementation outcomes will be adoption and fidelity evaluation of the digital peer support training curriculum, the feasibility and acceptability of Acceset in providing continuous access to online peer support throughout the duration of the seekers' engagement. The clinical outcomes will include Mattering, self-hood, compassion, mindfulness, psychological well-being scores for befrienders and seekers, and additionally perceived social support for seekers. The mechanism of change linking befrienders' support and seekers' mental well-being will be assessed using latent growth curve modelling.

Data Collection, Management and Analyses: We conducted power analysis to ascertain the adequate sample size needed for the randomized controlled trial, specifically in comparing the intervention and control groups on different clinical outcomes, so that the study has sufficient power to detect valid effects. The study sample size of n = 50 for intervention and n = 50 for control is needed because of multiple dependent variables measuring clinical outcomes included in the study and the testing of implementation outcomes (i.e., feasibility, utility). In dealing with missing data, we will first determine if missing data is missing completely at random (MCAR). If missing data is not systematic, as indicated by the non-significant result from Little's Missing Completely at Random Test, this study will handle missing data using full information maximum likelihood imputation.

Data will be analyzed and interpreted through three means. First, independent sample t-tests will be conducted whenever we need to compare intervention vs. control group on the different clinical outcomes in this study. Second, to elucidate the content of emotional disclosure on the Acceset platform, particularly in relation to the four active ingredients of psychological well-being (i.e., Mattering, self-hood, compassion and mindfulness), we will perform topic modelling using Latent Dirichlet Allocation (LDA) analyses with R to filter the huge amount of data available and drill down relevant themes and topics. LDA is an advanced statistical method that increases precision and accuracy in coding as compared to the exclusive use of qualitative approach /analyses. Third, to compare the mechanism of change , we will use Latent Growth Curve Modelling (LCM) to examine the trajectories of Acceset intervention in predicting the change in clinical outcomes experienced by youths. LCM elucidates whether an increasing trend in befrienders' digital peer support predicts increasing trends in youths' sense of Mattering, self-hood, compassion, mindfulness, and psychological well-being (i.e., clinical outcomes).

ELIGIBILITY:
Inclusion Criteria:

* youths aged 19 to 25 selective (distressed but healthy)
* primary indicative (exhibiting some symptoms but can't formally diagnose for anxiety, /depression or mental health disorder).

Exclusion Criteria:

--youths with high risk for suicidality detected at the time of screening with a validated psychological scale-PHQ-9.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Change in anxiety scores across 4 time points (seekers, befrienders): baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects) | baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects)
  Anxiety; 7-item General Anxiety Disorder Questionnaire; Self-reported measure; score range: 0 to 3, with higher score indicating greater anxiety severity Spitzer RL, Kroenke K, Williams JB, Löwe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of internal medicine 2006 May 22;166(10):1092-7.
Change in depression scores across 4 time points (seekers, befrienders): baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects) | baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects)
  Depression; 9-item Patient Health Questionnaire; Self-reported measure; score range: 0 to 3, with higher scores reflecting greater depression severity Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. Journal of General Internal Medicine 2001 Sep; 16(9):606-13. [doi: 10.1046/j.1525-1497.2001.016009606.x]

SECONDARY OUTCOMES:
Active ingredients of youth mental well-being (befrienders)--Mattering | Immediately before the start of digital peer support training and right after the training ends
  Content or qualitative analysis of befrienders' responses using the Rosenberg Mattering scale; score range: 1 to 4, with higher score indicating greater sense of mattering.
  Rosenberg, M., & McCullough, B. C. (1981). Mattering: Inferred significance and mental health among adolescents. Research in Community & Mental Health, 2, 163-182.
Active ingredients of youth mental well-being (befrienders)--self-hood, | Immediately before the start of digital peer support training and right after the training ends
  Content or qualitative analysis of befrienders' responses using three sub-scales on Self-knowledge: the internal self in you that reflects on things on hindsight Interpersonal self: how our self evolves based on who we are with Self as agent: the self that you build up based on the choices you make to achieve a future target score range: 1 to 4, with higher score indicating stronger self-hood
  Baumeister, R. F. (2010). The self. In R. F. Baumeister & E. J. Finkel (Eds.), Advanced social psychology: The state of the science (pp. 139-175). Oxford University Press.)
Active ingredients of youth mental well-being (befrienders)--compassion | Immediately before the start of digital peer support training and right after the training ends
  Content or qualitative analysis of befrienders' responses using the Fears of Compassion Scales. Score range: 0 to 4, lower scores indicate greater compassion (i.e., decreased fear of compassion).
  Self-Compassion Scale (SCS; Neff 2003). score range: 1 to 5, with higher score indicating higher compassion
  Gilbert, P., McEwan, K., Matos, M., & Rivis, A. (2010). Fears of compassion: Development of three selfreport measures. Psychology and Psycotherapy: Theory, Research and Practice. doi: 10.1348/147608310X526511.
  Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250. doi:10.1080/15298860309027.
Active ingredients of youth mental well-being (befrienders)--mindfulness | Immediately before the start of digital peer support training and right after the training ends
  Content or qualitative analysis of befrienders' responses using the mindfulness subscale from the Self-Compassion Scale (SCS; Neff 2003a). score range: 1 to 5, with higher score indicating higher mindfulness
  Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250. doi:10.1080/15298860309027.
Change in College adjustment scores across 4 time points (seekers, befrienders): baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects) | baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects)
  Student Adaptation to College Questionnaire; Self-reported measure; score range: 1 to 9, with higher score indicating better adjustment.
  Baker RW, Siryk B. Measuring adjustment to college. Journal of counseling psychology 1984 Apr;31(2):179.
Change in perceived social support across 4 time points (seekers): baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects) | baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects)
  Multidimensional Scale of Perceived Social Support (MSPSS); Self-reported measure; score range: 1 to 7, with higher score indicating greater perceived social support.
  Zimet GD Dahlem N Zimet SG Farley GK 1994 The Multidimensional Scale of Perceived Social Support (MSPSS) In J. F.Kevin (Ed.) The measures for clinical practice: A sourcebook Vol 2 Adults(2nd ed.) New York The Free Press
Change in Mattering scores across 4 time points (seekers, befrienders): baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects) | baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects)
  Rosenberg Mattering scale; Self-reported measure; score range: 1 to 4, with higher score indicating greater sense of mattering.
  Rosenberg, M., & McCullough, B. C. (1981). Mattering: Inferred significance and mental health among adolescents. Research in Community & Mental Health, 2, 163-182.
Client Satisfaction (seekers) | 3 weeks (the end of the intervention)
  Client Satisfaction Questionnaire (CSQ-8); Self-reported measure, score range: 1 to 4, with higher score indicating greater satisfaction Attkisson, C. C., & Greenfield, T. K. (2004). The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment: Instruments for adults (pp. 799-811). Lawrence Erlbaum Associates Publishers.
Client Satisfaction (befriender; digital peer support training program) | immediately after digital peer support training workshop
  Client Satisfaction Questionnaire (CSQ-8); Self-reported measure, score range: 1 to 4, with higher score indicating greater satisfaction Attkisson, C. C., & Greenfield, T. K. (2004). The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment: Instruments for adults (pp. 799-811). Lawrence Erlbaum Associates Publishers.
Focus group interview to assess barriers and facilitators of implementation and clinical effectiveness (befrienders, moderators) | 3 weeks (the end of the intervention)
  i. In assessing IMPLEMENTATION outcomes (i.e., whether Acceset intervention is feasible and acceptable), we will discuss with befrienders and moderators the following:
  1. Whether Acceset acts as a timely intervention i.e., in supporting youth seekers when they needed peer support? 2. Whether using Acceset is acceptable and satisfactory in terms of befrienders' attitudes towards the use of Acceset as an intervention (e.g., "I found Acceset easy to use")? ii. In assessing CLINICAL outcomes (i.e., whether Acceset improves or impacts positively the mental health outcomes), we will discuss with befrienders and moderators the following:
  1. Meaningful Aspect of Health: Whether and how Acceset supports youth seekers in their emotion management.
  2. Concept of Interest: Whether and how Acceset practically measures specific elements of emotion management using the emotion sticker pack.
  3. Endpoints: Whether and how Acceset captures precisely data that reflects outcomes of interest.
Change in Giving social support scores across 4 time points (befrienders): baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects). | baseline (before the intervention), 3 weeks (the end of the intervention), 6 weeks and 9 weeks (to measure carry over effects)
  Giving instrumental support to others (GISO); Self-reported measure, score range: Yes or No, with more Yes indicating a greater extent of giving instrumental support.
  Brown SL, Nesse RM, Vinokur AD, Smith DM. Providing social support may be more beneficial than receiving it: Results from a prospective study of mortality. Psychological Science 2003 Jul;14(4):320-7.
Burnout (befrienders) | 3 weeks (the end of the intervention)
  Oldenburg Burnout Inventory; Self-reported measure, score range: 1 to 4, with higher score indicating greater extent of burnout.
  Demerouti E, Mostert K, Bakker AB. Burnout and work engagement: a thorough investigation of the independency of both constructs. Journal of Occupational Health Psychology 2010 Jul;15(3):209.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Ho, PhD, Principal Investigator — N.1 Institute for Health, National University of Singapore; GeckHong Yeo, PhD, Study Director — N.1 Institute for Health, National University of Singapore
Locations (1):
- N.1 Institute for Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in article publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose-for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Marshall SK, Tilton-Weaver L. Adolescents' perceived mattering to parents and friends: Testing cross-lagged associations with psychosocial well-being. Int J Behav Dev 2019;43:541-52.
- [Background] Flett GL, Zangeneh M. Mattering as a vital support for people during the COVID-19 pandemic: The benefits of feeling and knowing that someone cares during times of crisis. J Concurr Disord 2020;2:106-23.
- [Background] Elliott G, Kao S, Grant A-M. Mattering: Empirical validation of a social-psychological concept. Self Identity 2004;3:339-54.
- [Background] Flett G, Khan A, Su C. Mattering and psychological well-being in college and university students: Review and recommendations for campus-based initiatives. Int J Ment Health Addict 2019;17:667-80.
- [Background] Flett GL, Nepon T. Mattering versus self-esteem in university students: associations with regulatory focus, social feedback, and psychological distress. J Psychoeduc Assess 2020;38:663-74.
- [Background] Joeng JR, Turner SL. Mediators between self-criticism and depression: Fear of compassion, self-compassion, and importance to others. J Couns Psychol. 2015 Jul;62(3):453-463. doi: 10.1037/cou0000071. Epub 2015 Mar 23. PMID 25798874
- [Background] Marshall SK. Do I matter? Construct validation of adolescents' perceived mattering to parents and friends. J Adolesc. 2001 Aug;24(4):473-90. doi: 10.1006/jado.2001.0384. PMID 11549327
- [Background] Rayle AD, Chung KY. Revisiting first-year college students' mattering: Social support, academic stress, and the mattering experience. J Coll Student Retent Res Theory Pract 2007;9:21-37.
- [Background] Marshall SK. Relative contributions of perceived mattering to parents and friends in predicting adolescents' psychological well-being. Percept Mot Skills. 2004 Oct;99(2):591-601. doi: 10.2466/pms.99.2.591-601. PMID 15560349
- [Background] Taylor J, Turner RJ. A longitudinal study of the role and significance of mattering to others for depressive symptoms. J Health Soc Behav. 2001 Sep;42(3):310-25. PMID 11668776
- [Background] Demir M, Davidson I. Toward a better understanding of the relationship between friendship and happiness: Perceived responses to capitalization attempts, feelings of mattering, and satisfaction of basic psychological needs in same-sex best friendships as predictors of happines. J Happiness Stud 2013;14:525-50.
- [Background] Dixon SK, Kurpius SER. Depression and college stress among university undergraduates: Do mattering and self-esteem make a difference? J Coll Stud Dev 2008;49:412-24.
- [Background] Flett GL, Su C, Ma L, et al. Mattering as a unique resilience factor in Chinese children: A comparative analysis of predictors of depression. Int J Child Adolesc Resil 2016;4:91-102.
- [Background] Flett GL, Burdo R, Nepon T. Mattering, insecure attachment, rumination, and self-criticism in distress among university students. Int J Ment Health Addict 2020.
- [Background] Baumeister RF. Self-concept, self-esteem, and identity. Personal. Contemp. theory Res., 1999, p. 339-75.
- [Background] Matera C, Bosco N, Meringolo P. Perceived mattering to family and friends, self-esteem, and well-being. Psychol Health Med. 2020 Jun;25(5):550-558. doi: 10.1080/13548506.2019.1626454. Epub 2019 Jun 3. PMID 31155928
- [Background] Demir M, Özen A, Doğan A, et al. I matter to my friend, therefore I am happy: Friendship, mattering, and happiness. J Happiness Stud 2011;12:983-1005.
- [Background] Demir M, Ozen A, Dogan A. Friendship, perceived mattering and happiness: a study of American and Turkish college students. J Soc Psychol. 2012 Sep-Oct;152(5):659-64. doi: 10.1080/00224545.2011.650237. PMID 22931003
- [Background] Vohs KD, Baumeister RF. Handbook of self-regulation: Research, theory, and applications. 2016.
- [Background] Wilson K. Can self-compassion reduce depression and anxiety in adolescents? Intuit BYU Undergrad J Psychol 2017;12:169-79.
- [Background] Chen-Bouck L, Patterson MM. Contingent self-worth in Chinese adolescents and young adults: Relations with global self-esteem and depressive symptoms. Soc Dev 2016;25:846-65.
- [Background] Gill C, Watson L, Williams C, Chan SWY. Social anxiety and self-compassion in adolescents. J Adolesc. 2018 Dec;69:163-174. doi: 10.1016/j.adolescence.2018.10.004. Epub 2018 Oct 13. PMID 30326397
- [Background] Masselink M, Van Roekel E, Oldehinkel AJ. Self-esteem in Early Adolescence as Predictor of Depressive Symptoms in Late Adolescence and Early Adulthood: The Mediating Role of Motivational and Social Factors. J Youth Adolesc. 2018 May;47(5):932-946. doi: 10.1007/s10964-017-0727-z. Epub 2017 Aug 7. PMID 28785953
- [Background] Orchard F, Pass L, Reynolds S. 'I Am Worthless and Kind'; the specificity of positive and negative self-evaluation in adolescent depression. Br J Clin Psychol. 2019 Sep;58(3):260-273. doi: 10.1111/bjc.12215. Epub 2018 Dec 16. PMID 30556150
- [Background] Raque-Bogdan TL, Ericson SK, Jackson J, Martin HM, Bryan NA. Attachment and mental and physical health: self-compassion and mattering as mediators. J Couns Psychol. 2011 Apr;58(2):272-278. doi: 10.1037/a0023041. PMID 21463033
- [Background] Cha M. The mediation effect of mattering and self-esteem in the relationship between socially prescribed perfectionism and depression: Based on the social disconnection model. Pers Individ Dif 2016;88:148-59.
- [Background] Nash SP, Longmore MA, Manning WD, Giordano PC. Strained Dating Relationships, A Sense of Mattering and Emerging Adults' Depressive Symptoms. J Depress Anxiety. 2015;Suppl 1:013. doi: 10.4172/2167-1044.S1-013. Epub 2015 Jun 18. PMID 26380799
- [Background] Bluth K, Campo RA, Futch WS, Gaylord SA. Age and Gender Differences in the Associations of Self-Compassion and Emotional Well-being in A Large Adolescent Sample. J Youth Adolesc. 2017 Apr;46(4):840-853. doi: 10.1007/s10964-016-0567-2. Epub 2016 Sep 15. PMID 27632177
- [Background] Lattie EG, Adkins EC, Winquist N, Stiles-Shields C, Wafford QE, Graham AK. Digital Mental Health Interventions for Depression, Anxiety, and Enhancement of Psychological Well-Being Among College Students: Systematic Review. J Med Internet Res. 2019 Jul 22;21(7):e12869. doi: 10.2196/12869. PMID 31333198
- [Background] Ali K, Farrer L, Gulliver A, Griffiths KM. Online Peer-to-Peer Support for Young People With Mental Health Problems: A Systematic Review. JMIR Ment Health. 2015 May 19;2(2):e19. doi: 10.2196/mental.4418. eCollection 2015 Apr-Jun. PMID 26543923
- [Background] Kaess M, Moessner M, Koenig J, Lustig S, Bonnet S, Becker K, Eschenbeck H, Rummel-Kluge C, Thomasius R, Bauer S; ProHEAD Consortium. Editorial Perspective: A plea for the sustained implementation of digital interventions for young people with mental health problems in the light of the COVID-19 pandemic. J Child Psychol Psychiatry. 2021 Jul;62(7):916-918. doi: 10.1111/jcpp.13317. Epub 2020 Sep 14. PMID 32924134
- [Background] Arnett JJ, Zukauskiene R, Sugimura K. The new life stage of emerging adulthood at ages 18-29 years: implications for mental health. Lancet Psychiatry. 2014 Dec;1(7):569-76. doi: 10.1016/S2215-0366(14)00080-7. Epub 2014 Dec 3. PMID 26361316
- [Background] Huckins JF, daSilva AW, Wang W, Hedlund E, Rogers C, Nepal SK, Wu J, Obuchi M, Murphy EI, Meyer ML, Wagner DD, Holtzheimer PE, Campbell AT. Mental Health and Behavior of College Students During the Early Phases of the COVID-19 Pandemic: Longitudinal Smartphone and Ecological Momentary Assessment Study. J Med Internet Res. 2020 Jun 17;22(6):e20185. doi: 10.2196/20185. PMID 32519963
- [Background] Shanahan L, Steinhoff A, Bechtiger L, Murray AL, Nivette A, Hepp U, Ribeaud D, Eisner M. Emotional distress in young adults during the COVID-19 pandemic: evidence of risk and resilience from a longitudinal cohort study. Psychol Med. 2022 Apr;52(5):824-833. doi: 10.1017/S003329172000241X. Epub 2020 Jun 23. PMID 32571438
- [Background] Rime, B. (2009). Emotion elicits the social sharing of emotion: Theory and empirical review. Emotion Review, 1, 60-85. https://doi.org/10.1177/1754073908097189
- [Background] Magson NR, Freeman JYA, Rapee RM, Richardson CE, Oar EL, Fardouly J. Risk and Protective Factors for Prospective Changes in Adolescent Mental Health during the COVID-19 Pandemic. J Youth Adolesc. 2021 Jan;50(1):44-57. doi: 10.1007/s10964-020-01332-9. Epub 2020 Oct 27. PMID 33108542
- [Background] Loades ME, Chatburn E, Higson-Sweeney N, Reynolds S, Shafran R, Brigden A, Linney C, McManus MN, Borwick C, Crawley E. Rapid Systematic Review: The Impact of Social Isolation and Loneliness on the Mental Health of Children and Adolescents in the Context of COVID-19. J Am Acad Child Adolesc Psychiatry. 2020 Nov;59(11):1218-1239.e3. doi: 10.1016/j.jaac.2020.05.009. Epub 2020 Jun 3. PMID 32504808
- [Background] Lippke S, Fischer MA, Ratz T. Physical Activity, Loneliness, and Meaning of Friendship in Young Individuals - A Mixed-Methods Investigation Prior to and During the COVID-19 Pandemic With Three Cross-Sectional Studies. Front Psychol. 2021 Feb 2;12:617267. doi: 10.3389/fpsyg.2021.617267. eCollection 2021. PMID 33603702
- [Background] Heimlich. (2012, December 14). Texting is nearly universal among young adult cell phone owners. https://www.pewresearch.org/fact-tank/2012/12/14/texting-is-nearly-universal-among-young-adult-cell-phone-owners/
- [Background] Liu, D., & Yang, C. C. (2016). Media niche of electronic communication channels in friendship: A meta-analysis. Journal of Computer-Mediated Communication, 21, 451-466. https://doi.org/10.1111/jcc4.12175
- [Background] Rimé, B. (2016). Self-disclosure. In H. S. Friedman (Ed.), Encyclopedia of mental health (pp. 66-74). MA: Academic Press. http://doi:10.1016/B978-0-12-397045-9.00075-6
- [Background] Choi, M., & Toma, C. L. (2014). Social sharing through interpersonal media: Patterns and effects on emotional well-being. Computers in Human Behavior, 36, 530-541. http://dx.doi.org/10.1016/j.chb.2014.04.026
- [Background] Marques de Miranda D, da Silva Athanasio B, Sena Oliveira AC, Simoes-E-Silva AC. How is COVID-19 pandemic impacting mental health of children and adolescents? Int J Disaster Risk Reduct. 2020 Dec;51:101845. doi: 10.1016/j.ijdrr.2020.101845. Epub 2020 Sep 10. PMID 32929399
- [Background] Nearchou F, Flinn C, Niland R, Subramaniam SS, Hennessy E. Exploring the Impact of COVID-19 on Mental Health Outcomes in Children and Adolescents: A Systematic Review. Int J Environ Res Public Health. 2020 Nov 16;17(22):8479. doi: 10.3390/ijerph17228479. PMID 33207689
- [Background] Bernecker SL, Williams JJ, Caporale-Berkowitz NA, Wasil AR, Constantino MJ. Nonprofessional Peer Support to Improve Mental Health: Randomized Trial of a Scalable Web-Based Peer Counseling Course. J Med Internet Res. 2020 Sep 21;22(9):e17164. doi: 10.2196/17164. PMID 32955451
- [Background] Kaylor-Hughes CJ, Rawsthorne M, Coulson NS, Simpson S, Simons L, Guo B, James M, Moran P, Simpson J, Hollis C, Avery AJ, Tata LJ, Williams L; REBOOT Notts Lived Experience Advisory Panel; Morriss RK. Direct to Public Peer Support and e-Therapy Program Versus Information to Aid Self-Management of Depression and Anxiety: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Dec 18;6(12):e231. doi: 10.2196/resprot.8061. PMID 29254909
- [Background] Myers AL, Collins-Pisano C, Ferron JC, Fortuna KL. Feasibility and Preliminary Effectiveness of a Peer-Developed and Virtually Delivered Community Mental Health Training Program (Emotional CPR): Pre-Post Study. J Particip Med. 2021 Mar 4;13(1):e25867. doi: 10.2196/25867. PMID 33661129
- [Background] Freeman E, Barker C, Pistrang N. Outcome of an online mutual support group for college students with psychological problems. Cyberpsychol Behav. 2008 Oct;11(5):591-3. doi: 10.1089/cpb.2007.0133. PMID 18817485
- [Background] Horgan A, McCarthy G, Sweeney J. An evaluation of an online peer support forum for university students with depressive symptoms. Arch Psychiatr Nurs. 2013 Apr;27(2):84-9. doi: 10.1016/j.apnu.2012.12.005. Epub 2013 Feb 13. PMID 23540518
- [Background] Andalibi N, Flood MK. Considerations in Designing Digital Peer Support for Mental Health: Interview Study Among Users of a Digital Support System (Buddy Project). JMIR Ment Health. 2021 Jan 4;8(1):e21819. doi: 10.2196/21819. PMID 33393909
- [Background] Fortuna KL, Naslund JA, LaCroix JM, Bianco CL, Brooks JM, Zisman-Ilani Y, Muralidharan A, Deegan P. Digital Peer Support Mental Health Interventions for People With a Lived Experience of a Serious Mental Illness: Systematic Review. JMIR Ment Health. 2020 Apr 3;7(4):e16460. doi: 10.2196/16460. PMID 32243256
- [Background] Flett, G. L., & Zangeneh, M. (2020). Mattering as a vital support for people during the COVID-19 pandemic: the benefits of feeling and knowing that someone cares during times of crisis. Journal of Concurrent Disorders, 2(1), 106-123.
- [Background] Rossi A, Panzeri A, Pietrabissa G, Manzoni GM, Castelnuovo G, Mannarini S. The Anxiety-Buffer Hypothesis in the Time of COVID-19: When Self-Esteem Protects From the Impact of Loneliness and Fear on Anxiety and Depression. Front Psychol. 2020 Nov 10;11:2177. doi: 10.3389/fpsyg.2020.02177. eCollection 2020. PMID 33240140
- [Background] Gonzalez-Garcia M, Alvarez JC, Perez EZ, Fernandez-Carriba S, Lopez JG. Feasibility of a Brief Online Mindfulness and Compassion-Based Intervention to Promote Mental Health Among University Students During the COVID-19 Pandemic. Mindfulness (N Y). 2021;12(7):1685-1695. doi: 10.1007/s12671-021-01632-6. Epub 2021 May 17. PMID 34025814
- [Background] Howard JL, Bureau J, Guay F, Chong JXY, Ryan RM. Student Motivation and Associated Outcomes: A Meta-Analysis From Self-Determination Theory. Perspect Psychol Sci. 2021 Nov;16(6):1300-1323. doi: 10.1177/1745691620966789. Epub 2021 Feb 16. PMID 33593153
- [Background] Levesque, R. J. R. (2011). Externalizing and internalizing symptoms. In R. J. R Levesque (Eds.), Encyclopedia of Adolescence (pp. 903-905). Springer Science & Business Media
- [Derived] Yeo G, Loo G, Oon M, Pang R, Ho D. A Digital Peer Support Platform to Translate Online Peer Support for Emerging Adult Mental Well-being: Randomized Controlled Trial. JMIR Ment Health. 2023 Apr 18;10:e43956. doi: 10.2196/43956. PMID 36756843
- [Derived] Yeo G, Chang W, Lee LN, Oon M, Ho D. A Digital Peer Support Platform to Translate Web-Based Peer Support for Emerging Adult Mental Well-being: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 20;11(9):e34602. doi: 10.2196/34602. PMID 36125855